CLINICAL TRIAL: NCT05459623
Title: Effects of Myofascial Release With and Without EMMETT Technique in Iliotibial Band Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR/20/1066 Faiza Altaf
Record Dates: First submitted 2021-05-03; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Iliotibial Band Syndrome
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual myofascial release (Active Comparator): Manual myofascial release as conventional treatment
  Interventions: Other: Manual myofascial release
- Emmett intervention (Experimental): Emmett intervention and myofascial release
  Interventions: Other: Emmett intervention

INTERVENTIONS:
Other: Manual myofascial release — will receive Manual myofascial release to iliotibial band by having the subject to lie in the side lying position on the unaffected side. The upper leg to be tested was rested on the table with hip and knee flexion. Then the therapist applied a few kilograms of force weight along the iliotibial band course proximally to distally. The therapist will repeat this for 6 minutes.
  Other Names: Group A
  Arms: Manual myofascial release
Other: Emmett intervention — will receive manual myofascial release and the Emmett intervention with the subject sitting upright on a 45cm wooden chair; light, constant pressure via the middle finger (at a perpendicular angle to the skin) will be applied at both points, three times for 10-20s with 5-10s breaks between. A light sweeping action over the sensory area that will treated will be performed once, using the back of the fingers. The rationale for this is that the light brushing action "disperses the sensory awareness to move without being too heavy or specific enough to create muscular response." The sequence performed on one side will then repeated on the opposite leg. In Ross Emmett's teachings of the technique he insists on treatment of both sides when focusing on the lower body (for balance). Once both sides will be completed, the subject will be instructed to walk around the room for a minute.
  Other Names: Group B
  Arms: Emmett intervention

SUMMARY:
The iliotibial (IT) tract or band is a lateral thickening of the fascia lata that is composed of the distal fusion of the muscular fascia of the gluteus maximus and tensor fascia lata muscles. The iliotibial tract travels along the lateral side of the thigh and across the knee joint, inserting on the lateral epicondyle of the tibia. A tight IT band has been diagnosed in several problems related to the knee including patellofemoral syndrome and iliotibial band syndrome. Several authors have suggested that tightness in the IT band may contribute to patellofemoral syndrome and knee pain by pulling the patella laterally thereby causing abnormal tracking of the patella in the trochlear groove. Stretching of the iliotibial band is frequently recommended in treatment programs for patients with LBP. Because the iliotibial band attaches to the ilium, tightness of this muscle is thought to cause anterior innominate rotation and lateral pelvic tilt. The Ober test is performed to assess tightness in the iliotibial band.

The term myofascial release encompasses various techniques used to release fascial restrictions. Many forms of bodywork that includes a soft tissue technique exist with Bowen therapy, Emmett technique, deep tissue massage, neuromuscular techniques (NMT), Muscle Energy Techniques (MET) and foam rolling.

This study focusses on effects of myofascial release with Emmett technique. This study will be conducted in a clinical set up (Saba's physical therapy, rehabilitation and sports injury clinic in Gulberg 3) and will take 6 months. Study will be conducted on 22 subjects involving 11 subjects in each group. Group A will be given myofascial release only and group B will be given myofascial release with Emmett technique. Total duration of study will be three weeks and assessment will be done before treatment and after every week. Numeric pain rating scale, goniometer and vertical jump test are used for assessing pain, flexibility and power respectively.

ELIGIBILITY:
Inclusion Criteria:

* Positive Ober's Test
* Both males and females
* Age 25 to 45 years

Exclusion Criteria:

* TFL (Tensor Fascia Lata) tightness
* Any pathological and traumatic conditions, Fractures and Dislocation,
* Already received few sessions of Manual Therapy treatment
* Taking corticosteroids, analgesic or anti-inflammatory drugs.
* Treatment of lower limb myofascial pain or trigger points at the time of the study • Current or previous symptoms of pathology reported in the lower limbs or pelvis

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 2 months
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Range of Motion | 2 months
  Standard Goniometer was used to measure how far you can move or stretch a part of your body, such as a joint or a muscle specifically hip joint
Vertical Jump test | 2 Months
  The Vertical Jump test is designed to measure an applicants lower body strength in . The test is conducted using a vertical jump test gauge. Height was measured in inches or cm The mechanical work performed to accomplish a vertical jump can be determined by using the jump height distance that was measured (using Work = Force x Distance where Force = Mass x Acceleration).

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah IU, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fairclough J, Hayashi K, Toumi H, Lyons K, Bydder G, Phillips N, Best TM, Benjamin M. The functional anatomy of the iliotibial band during flexion and extension of the knee: implications for understanding iliotibial band syndrome. J Anat. 2006 Mar;208(3):309-16. doi: 10.1111/j.1469-7580.2006.00531.x. PMID 16533314
- [Background] Hudson Z, Darthuy E. Iliotibial band tightness and patellofemoral pain syndrome: a case-control study. Man Ther. 2009 Apr;14(2):147-51. doi: 10.1016/j.math.2007.12.009. Epub 2008 Mar 3. PMID 18313972
- [Background] Reese NB, Bandy WD. Use of an inclinometer to measure flexibility of the iliotibial band using the Ober test and the modified Ober test: differences in magnitude and reliability of measurements. J Orthop Sports Phys Ther. 2003 Jun;33(6):326-30. doi: 10.2519/jospt.2003.33.6.326. PMID 12839207
- [Background] Lavine R. Iliotibial band friction syndrome. Curr Rev Musculoskelet Med. 2010 Jul 20;3(1-4):18-22. doi: 10.1007/s12178-010-9061-8. PMID 21063495
- [Background] Okamoto T, Masuhara M, Ikuta K. Acute effects of self-myofascial release using a foam roller on arterial function. J Strength Cond Res. 2014 Jan;28(1):69-73. doi: 10.1519/JSC.0b013e31829480f5. PMID 23575360
- [Background] Bevilaqua-Grossi D, Monteiro-Pedro V, Sousa G, Silva Z, Bérzin F. Contribution to the anatomical study of the oblique portion of the vastus lateralis muscle. Braz J Morphol Sci. 2004;21(1):47-52.
- [Background] Ercole B, Antonio S, Julie Ann D, Stecco C. How much time is required to modify a fascial fibrosis? J Bodyw Mov Ther. 2010 Oct;14(4):318-25. doi: 10.1016/j.jbmt.2010.04.006. Epub 2010 May 20. PMID 20850038